CLINICAL TRIAL: NCT03877445
Title: Study of the Influence of Blue Light Emitted by Computer / Television Screens on Melasma Single-center, Interventional, Randomized, Single-blind Study (Masked Investigator) MELABLUE Study
Brief Title: Study of the Influence of Blue Light Emitted by Computer / Television Screens on Melasma MELABLUE Study
Acronym: MELABLUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 19-PP-02
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melasma Group exposed left half-face by ORIEL solar simulator (Other): Twelve patients will be included in the study and exposed on a half-face from Day1 to Day5. The other half-face will serve as unexposed control.
  Interventions: Device: exposition half-face
- Melasma Group exposed right half-face by ORIEL solar simulator (Other): Twelve patients will be included in the study and exposed on a half-face from Day1 to Day5. The other half-face will serve as unexposed control.
  Interventions: Device: exposition half-face

INTERVENTIONS:
Device: exposition half-face — Patients will be included in the study and exposed on a half-face from Day1 to Day5. The other half-face will serve as unexposed control. The effect of blue light on the melasma lesions will be assessed from Day 1 to Day 6 using chromametry and a modified Melasma Area and Severity Index on standardized photographs

SUMMARY:
Melasma is a fairly common condition resulting in hyperpigmented macules on the face. Melasma is difficult to treat and has a significant negative impact on the patient's quality of life.

Melasma is worsen when exposed to high energy visible light (blue and violet light) of the solar spectrum. Blue light emitted by LED screens from computers, tablets, televisions and even mobile phones is currently suspected (via media channels) to induce harmful effects on the skin, including pigmentation and photoaging. These screens, however, emit much lower irradiances than those of the solar spectrum, and the probability that these irradiances impact the skin is very low.

The objective of the study is to assess the effect of blue light emitted by computer/television screens on the intensity of melasma pigmentation. To do this, it is proposed to use maximized conditions that could be encountered in normal daily life, namely a simulation of blue light exposure (420-490nm) at 20 cm from a laptop LED screen, 8 hours a day for 5 days. Since it is not proposed to expose a person for 8 hours a day, a solar simulator with appropriate filters will be used to emit a spectrum of between 420 and 490 nm with a compatible intensity for an acceptable duration of exposure (around 30 minutes a day).

Twelve patients will be included in the study and exposed on a half-face from Day1 to Day5. The other half-face will serve as unexposed control. The effect of blue light on the melasma lesions will be assessed from Day 1 to Day 6 using chromametry and a modified MASI on standardized photographs. A final evaluation visit will be performed at Day 15.

ELIGIBILITY:
Inclusion Criteria:

* Female patient, 18 years of age and older, phototype II to V on the Fitzpatrick scale
* Patient with a clinically diagnosed diagnosis of melasma.
* Patient without a serious medical history and declared fit to participate in the medical visit.
* Patient who has signed a written informed consent form before any action related to the study is initiated.
* If the patient is able to procreate, she should use reliable contraception (contraceptive pill, contraceptive implant, intrauterine contraceptive device, bilateral tubal ligation / section, condoms), and agree not to change contraceptive status for at least one month before the start of the study and throughout the duration of the study.

Exclusion Criteria:

* Women who are pregnant or breastfeeding or who have planned a pregnancy during the course of the study.
* Patient with another pigment condition on the face.
* Patient who used depigmenting cosmetic on the face in the two weeks prior to inclusion.
* Patient who used a local corticosteroid on the face or systemic steroids during the month prior to inclusion.
* Patient who used local tretinoin or local hydroquinone during the month prior to inclusion.
* Patient who took systemic or topical photosensitizing treatments during the month preceding the first day of the study (1 month or 5 half-lives, the longest possible duration),
* Patient with a history of photodermatoses.
* Patient spending more than 3 hours a day in front of a screen (computer, LED TV, tablet, phone etc ...) for professional or private reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of blue light emitted by computer / television screens on the intensity of pigmentation of melasma by Melasma Area and Severity Index scale | 15 days

SECONDARY OUTCOMES:
Evaluate the tolerance and the possible undesirable effects induced by the exposure in blue light with Melasma Area and Severity Index scale | 15 days
Evaluate the effect of blue light emitted by computer / television screens on the intensity of pigmentation of healthy skin by chomametry | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PASSERON, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Centre de Pharmacologie Clinique Appliquée à la Dermatologie, Nice, France